CLINICAL TRIAL: NCT01050387
Title: A Randomized, Controlled Trial of Vitamin D Supplementation in Infants and Children: Effects of Vitamin D Dose and Genotype of the Binding Protein
Brief Title: Effects of Vitamin D Dose and Genotype of the Binding Protein in Infants and Children
Acronym: VitaD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Thrasher Research Fund (Other)
Responsible Party: Principal Investigator, Thomas Carpenter, Professor, Yale University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0909005699; 1RC1HD063562 (NIH); M#136410
Record Dates: First submitted 2010-01-13; First posted 2010-01-15 (Estimated); Last update posted 2014-08-05 (Estimated); Status verified 2013-07

CONDITIONS: Vitamin D Deficiency
Keywords: Vitamin D Deficiency; VDD; Vitamin D Supplementation; Vitamin D Binding Protein; DBP; Nutritional rickets; rickets; 25hydroxyvitamin D; 25OHD; 1,25OH2D; vitamin D metabolites; PTH; vitamin D homeostasis
MeSH Terms: conditions — Vitamin D Deficiency; Rickets | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Dietary Supplement: Vitamin D — Vitamin D (either 400 IU vs 1000 IU) given orally each day

SUMMARY:
The purpose of this study is to determine if the vitamin D binding protein genotype influences circulating vitamin D levels and if it may have functional consequences on vitamin D activity.

DETAILED DESCRIPTION:
Vitamin D has recently been the subject of much attention. Advantages to the prevention of vitamin D deficiency (VDD) in young children are obvious: acutely, hypocalcemic seizures may occur in VDD, and rickets can result in long-term skeletal deformities. Previous research has emphasized the importance of identifying optimal supplementation doses and appropriate target thresholds for circulating 25-hydroxyvitamin D (25-OHD), the best described marker of vitamin D status. The timely next step is to objectively establish effective doses for the prevention of VDD, without creating risk from overzealous supplementation, in a population representative of those most at risk for overt disease.

Although the primary role of vitamin D is considered to be its effect on intestinal calcium absorption, enormous variability of fractional calcium absorption in relation to 25-OHD levels exists. We provide evidence that a significant component of this variability is genetic in nature and in particular, relates to vitamin D binding protein (DBP) genotype.

The aggregate data suggest that the critical mechanism for the development of nutritional rickets is reduction in availability of calcium to the skeleton, which is largely determined by vitamin D status and intestinal calcium absorption. Our proposal focuses on the establishment of a workable definition of vitamin D deficiency in an underserved and highly vulnerable population and to assess the impact of genetic variance in VDR and DBP as factors to be considered in the recommendation of vitamin D status assessment, taking into account the outcome of 25-OHD level, and in additional studies, potential functional consequences of vitamin D related to both its classical and non-classical effects.

ELIGIBILITY:
Inclusion Criteria:

* 6 months to 6 years of age
* healthy or free from any diseases or conditions that may affect nutritional status or bone metabolism
* willingness of family to participate in a 6-month study of vitamin D supplementation

Exclusion Criteria:

* Chronic disease
* Prematurity < 32 weeks gestational age
* Liver disease such as hepatitis or renal/urologic disease (e.g., recurrent urinary tract infection)
* Use of pharmacologic or prescription-level dosages of vitamin D or its metabolites. We will exclude users of any systemic glucocorticoid preparation and users of inhaled steroids that are considered greater than medium dose for age 4 yrs. Specifically, this would exclude users of over 1 mg/day of budesonide, and over 352 mcg/day of fluticasone.
* Current or recent (within 1 month) use of anticonvulsants or other medications known to affect bone and mineral homeostasis or alkaline phosphatase levels.

Ages: 6 Months to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 193 (Actual)
Dates: Start 2010-01; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Changes in serum 25-OH vitamin D | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Thomas O Carpenter, M.D., Principal Investigator — Yale University
Locations (1):
- Yale University School of Medicine, New Haven, Connecticut, United States

REFERENCES:
- [Background] Gungor N, Saad R, Janosky J, Arslanian S. Validation of surrogate estimates of insulin sensitivity and insulin secretion in children and adolescents. J Pediatr. 2004 Jan;144(1):47-55. doi: 10.1016/j.jpeds.2003.09.045. PMID 14722518
- [Background] DeLucia MC, Mitnick ME, Carpenter TO. Nutritional rickets with normal circulating 25-hydroxyvitamin D: a call for reexamining the role of dietary calcium intake in North American infants. J Clin Endocrinol Metab. 2003 Aug;88(8):3539-45. doi: 10.1210/jc.2002-021935. PMID 12915633
- [Background] Heaney RP, Davies KM, Chen TC, Holick MF, Barger-Lux MJ. Human serum 25-hydroxycholecalciferol response to extended oral dosing with cholecalciferol. Am J Clin Nutr. 2003 Jan;77(1):204-10. doi: 10.1093/ajcn/77.1.204. PMID 12499343
- [Background] Safadi FF, Thornton P, Magiera H, Hollis BW, Gentile M, Haddad JG, Liebhaber SA, Cooke NE. Osteopathy and resistance to vitamin D toxicity in mice null for vitamin D binding protein. J Clin Invest. 1999 Jan;103(2):239-51. doi: 10.1172/JCI5244. PMID 9916136
- [Background] Zella LA, Shevde NK, Hollis BW, Cooke NE, Pike JW. Vitamin D-binding protein influences total circulating levels of 1,25-dihydroxyvitamin D3 but does not directly modulate the bioactive levels of the hormone in vivo. Endocrinology. 2008 Jul;149(7):3656-67. doi: 10.1210/en.2008-0042. Epub 2008 Mar 27. PMID 18372326
- [Background] Pettifor JM. Nutritional Rickets. In: Pediatric Bone: Biology and Diseases. Glorieux FH, Pettifor JM, Juppner H (eds.) Academic Press: San Diego, CA, p 541-565, 2003.
- [Derived] Simpson CA, Zhang JH, Vanderschueren D, Fu L, Pennestri TC, Bouillon R, Cole DEC, Carpenter TO. Relationship of Total and Free 25-Hydroxyvitamin D to Biomarkers and Metabolic Indices in Healthy Children. J Clin Endocrinol Metab. 2020 Apr 1;105(4):e1631-40. doi: 10.1210/clinem/dgz230. PMID 31774125